CLINICAL TRIAL: NCT02398942
Title: A Prospective Study of Proximal Pole Fractures of the Scaphoid
Brief Title: Proximal Pole Fractures of the Scaphoid
Status: Withdrawn | Type: Observational
Why Stopped: The investigator left the institution so the study was terminated.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Medical Center Haaglanden, The Hague, The Netherlands (Unknown); Skane University Hospital (Other); Ghaem Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Chief of Orthopaedic Hand and Upper Extremity Service, Massachusetts General Hospital
Other Study IDs: 2015P000177
Record Dates: First submitted 2015-03-04; First posted 2015-03-26 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Proximal Pole Fractures of the Scaphoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Proximal Pole Fracture of the Scaphoid: QuickDASH 6 months after injury CT scan 6 months after injury

SUMMARY:
Aim:

The aim of this study is to analyze the clinical and radiological outcomes of patients with a proximal pole fracture of the scaphoid

Primary null hypothesis:

There are no factors associated with nonunion of a proximal pole fracture of the scaphoid.

Secondary null hypothesis:

Patients with an acute proximal pole fracture of the scaphoid have QuickDASH (Disabilities of the Arm, Shoulder, and Hand) scores at or above the population norm (a score of 13 in the Norway and 10.9 in the United States), 2 to 6 months after injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Proximal pole fracture of the scaphoid on computed tomography scans made in the planes defined by the long axis of the scaphoid. The proximal pole will be defined as the proximal fifth of the scaphoid, excluding small scapholunate ligament avulsion fractures.
* Interval between injury and diagnosis of less than 2 weeks.
* English or Spanish fluency and literacy

Exclusion Criteria:

* Pregnant women
* Inability to complete enrollment forms due to any mental status or language problems (e.g. dementia, head injury, overall illness).
* Patients with other fractures or injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with proximal pole fracture of the scaphoid
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Disability measured using QuickDASH | 6 months
Nonunion of Fracture | 6 months
  The nonunion of the fracture will be measured using CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD PhD, Principal Investigator — Massachusetts General Hospital